CLINICAL TRIAL: NCT05985018
Title: A Randomized Trial of Traditional Dietary Advice Versus Mediterranean Diet in Irritable Bowel Syndrome
Brief Title: Traditional Dietary Advice Vs. Mediterranean Diet in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH20655b
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Dietary Advice (Active Comparator): Its main elements are to adopt sensible eating habits and avoid excess fatty foods, spicy foods, processed foods, caffeine, fizzy drinks and alcohol.
  Interventions: Other: Traditional Diet
- Mediterranean Diet (Active Comparator): The principle components is a diet rich in vegetables, pulses, whole grains, and olive oil
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Traditional Diet — Provided as an educational leaflet
  Arms: Traditional Dietary Advice
Other: Mediterranean Diet — Provided as an educational leaflet
  Arms: Mediterranean Diet

SUMMARY:
Irritable bowel syndrome (IBS) affects 5-10% of the population, and incurs substantial health impairment and healthcare utilization. Over 80% of individuals with IBS report food to trigger or aggravate symptoms, with many seeking to undertake dietary modifications. Current guidelines recommend first-line therapy with the relatively straightforward traditional dietary advice, with the more complex and restrictive low FODMAP diet reserved as second-line therapy.

There is emerging data suggesting that the Mediterranean diet may also improve the symptoms of IBS, although it has not yet been subject to any head-to-head randomized dietary trials to help position it within the treatment algorithm. Given the relative ease of implementing the Mediterranean diet, alongside its recognized cardio-metabolic and mental health benefits, studying its efficacy in IBS is attractive as it could potentially pave the way for another first-line dietary option being available to patients before escalating to the demanding and resource intensive second-line therapies.

The investigators will perform a randomized trial comparing the clinical efficacy of traditional dietary advice vs. a Mediterranean diet in IBS. Following dietary randomization, participants will complete validated questionnaires to assess changes in IBS symptoms, quality of life, mood, somatic symptoms, nutritional status, as well as dietary satisfaction and adherence.

ELIGIBILITY:
Inclusion Criteria:

* IBS Symptom Severity Scale(IBS-SSS) > 75
* Online access
* English literate

Exclusion Criteria:

* Organic gastrointestinal diseases (e.g. inflammatory bowel disease, GI cancer, coeliac disease, microscopic colitis, bile acid diarrhoea)
* Major abdominal surgery (except laparoscopy, appendectomy, cholecystectomy)
* History of eating disorder
* Body mass index <20
* Current dietary interventions
* Current use of opioids/antibiotics
* Titrating dose of neuromodulators
* Severe systemic disease (e.g. cardiac, renal, respiratory, psychiatric) necessitating frequent medical consultations/hospitilisations
* Pregnant
* Diabetes mellitus
* Scleroderma
* Memory impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of IBS patients experiencing clinical response with traditional dietary advice vs. Mediterranean diet | Baseline to Week 6
  IBS symptom severity scale (IBS-SSS) where a 50-point reduction denotes a meaningful clinical response

SECONDARY OUTCOMES:
Changes in individual items of the IBS-SSS | Baseline to Week 6
  IBS- SSS contains 5 specific questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) with score ranging from 0-100. Change in individual items will be compared within- and between- groups.
Changes in Anxiety and Depression | Baseline to Week 6
  The four-item patient health questionnaire (PHQ-4) for anxiety and depression is a validated questionnaire assessing mood, with higher scores representing worse mood. Change in scores will be compared within- and between- groups
Changes in Somatic Symptom reporting | Baseline to Week 6
  The validated patient health questionnaire-12 assess extra-intestinal somatic symptoms, with higher scores representing greater somatic symptom severity. Change in scores will be compared within- and between- groups
Changes in quality of life | Baseline to Week 6
  The validated Short form 8 Quality of life Questionnaire assesses quality of life, with higher scores representing better quality of life. Change in scores will be compared within- and between- groups
Dietary satisfaction to assigned intervention | Week 6
  The Diet Satisfaction Score is a 10-item questionnaire assessing dietary satisfaction to an allocated diet (either Mediterranean diet or traditional diet), with higher scores representing greater satisfaction. Changes in score will be compared between the groups.
Adherence to the Mediterranean diet | Week 6
  The 14-point Mediterranean Diet Adherence Screener will check adequate dietary adherence, which we expect will be seen in those assigned a Mediterranean diet compared with traditional diet. Higher scores represent better adherence.
Changes in nutritional intake | Baseline to Week 6
  The Comprehensive Nutritional Assessment Questionnaire assesses macronutrient and micronutrient intake, FODMAPs, fibre, starch, glycaemic index/load. Change in scores will be compared within- and between- groups. Only a subset will complete this

CONTACTS AND LOCATIONS:
Overall Officials: Imran Aziz, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bamidele JO, Brownlow GM, Flack RM, Buckle RL, Shaw CC, Shiha MG, Aziz I. The Mediterranean Diet for Irritable Bowel Syndrome : A Randomized Clinical Trial. Ann Intern Med. 2025 Dec;178(12):1709-1717. doi: 10.7326/ANNALS-25-01519. Epub 2025 Oct 28. PMID 41144975